CLINICAL TRIAL: NCT01888055
Title: Influence of Transcranial Direct-current Stimulation on Cortical Plasticity in Healthy Older Adults
Brief Title: Influence of tDCS on Cortical Plasticity in Healthy Older Adults
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not funded
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Agnes Flöel, Prof. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Plasticity in healthy adults
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Healthy Older Adults
Keywords: Healthy older adults Cortical Plasticity; Transcranial Direct Current Stimulation
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- transcranial direct current stimulation (Experimental)
  Interventions: Device: transcranial direct current stimulation
- sham stimulation (Placebo Comparator)
  Interventions: Device: sham stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation
  Arms: transcranial direct current stimulation
Device: sham stimulation
  Arms: sham stimulation

SUMMARY:
The aim of this study is to investigate whether the anodal transcranial direct current stimulation (tDCS) over the primary motor cortex (M1) in healthy older adults leads to an increase in cortical plasticity (change in motor evoked potentials (MEP) in mV).

ELIGIBILITY:
Inclusion Criteria:

* right-handed according to the Oldfield Händigkeits inventory (lateralization index >70)(1971)
* no obvious cognitive impairment (MMSE>26, Demtect>13)
* age between 50 and 80 years

Exclusion Criteria:

* Severe neurological / psychiatric or pre-existing internist conditions because additional cognitive deficits are expected
* Epilepsy, epileptic seizure in medical history
* Cognitive deficit (MMSE <20)
* Depressive episode (Beck Depression Inventory (BDI) > 12)
* intake of centrally active drugs <3 months , particularly acetylcholinesterase inhibitors
* Pregnancy
* Pacemaker (contraindication for MRI)
* Other metal parts in the body (contraindication for MRI)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
anodal transcranial direct current stimulation (tDCS) over the primary motor cortex (M1) in healthy older adults | 1 week
  to investigate whether the anodal transcranial direct current stimulation over the primary motor cortex (M1) in healthy older adults increases cortical plasticity (measured via motor evoked potentials)compared to sham stimulation

SECONDARY OUTCOMES:
Comparison of tDCS-induced changes on central cholinergic activity | 1 week
  to investigate weather anodal transcranial direct-current stimulation affect central cholinergic activity (measured via a TMS-protocol) in healthy older adults compared to sham stimulation
Comparison of tDCS-induced changes in the learning success | 1 week
  tDCS-induced changes on learning success (performance in a motor learning paradigm in healthy older adults after tDCS vs. sham)
MR elastography | 1 week
  Comparison of viscoelastic parameters in cerebral MR elastography in healthy older adults
genetic polymorphism, ApoE4 | once
  optional assessment of genetic Apo4 epsilon status for assessment of differences in cortical plasticity and elasticity between Apo4 epsilon positive and negative participants

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik und Poliklinik für Neurologie, Charité Universitätsmedizin Berlin, Berlin, Germany